CLINICAL TRIAL: NCT02818062
Title: Severe Intraocular Infection
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 3964
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Endophthalmitis
Keywords: Endophthalmitis; Cytokines; Chemokines; Inflammation; Regulation
MeSH Terms: conditions — Endophthalmitis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humor obtained by anterior chamber tap.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endophthalmitis: The diagnosis of endophthalmitis was made on the basis of clinical features including pain, decreased visual acuity (VA), diffuse bulbar conjunctival hyperaemia, chemosis, inflammation of the anterior segment and posterior segment inflammation (all patients had vitreous infiltration diagnosed by biomicroscopy or ophthalmic ultrasound).
  Interventions: Biological: Cytokines dosage in Aqueous humor
- Cataract (Control): Controls were patients who underwent cataract surgery.
  Interventions: Biological: Cytokines dosage in Aqueous humor

INTERVENTIONS:
Biological: Cytokines dosage in Aqueous humor — Specify details not covered in associated Arm Description.

SUMMARY:
The host-immune reaction to infection is essential for the comprehension of the disease and the development of new therapies.

The aim of the study is to describe intraocular cytokines network in aqueous humor using multiplex immunoassay, during severe intraocular infection.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative endophthalmitis
* Cataract

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from referral centers coming for post-operative endophthalmitis. Multicenter studies (in France: Strasbourg, Dijon, Grenoble, Nancy).
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Intraocular cytokine network. Intraocular levels of 27 cytokines | Once in the 24 hours following the admission
  Cytokines and chemokines levels in Aqueous humor (AqH) are measured with the Bio-Plex® Multiplex System human Cytokine 27-Plex Panel assay (Bio-Rad, Marne-la-Coquette, France).
  The immune mediators were classified in five categories: (a) proinflammatory mediators: (IL-6 and monocyte chemoattractant protein (MCP-1), (b) type 1 cytokines: IL-2, IL-12(p70), Interferon (IFN-γ), and tumor necrosis factor-α (TNF-α), (c) type 2 cytokines: IL-4, IL-10 and IL-13, (d) T-regulatory cytokine: IL-10 and (e) Th-17 cytokine: IL-17. The cytokine and chemokine assay plate layout consisted of a standard series in duplicate (1 to 32 000 pg/ml), four blank wells and 20 μl duplicates of pooled AqH samples, diluted to 50 μl with BioPlex mouse serum diluent. The BioPlex® method was performed as recommended by the manufacturer and previously published studies. Data were analyzed with Bio-Plex Manager software® V 1.1 (Bio-Rad).

SECONDARY OUTCOMES:
Visual acuity | Once in the 24 hours following the admission, then 3 months, 6 months and 1 year
  E Snellen Conversion in LogMAR unit

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Service d'Ophtalmologie, Hôpital Pasteur, Colmar
  - Service d'Ophtalmologie, Hôpital Général de Dijon, Dijon
  - Service d'Ophtalmologie, Hôpital Michallon, Grenoble
  - Service d'Ophtalmologie, Centre Hospitalier de Mulhouse, Mulhouse
  - Service d'Ophtalmologie, CHU de Nancy, Nancy
  - Service d'Ophtalmologie, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service d'Ophtalmologie, Hôpital de Brabois, Vandœuvre-lès-Nancy